CLINICAL TRIAL: NCT05817370
Title: Integrated Model for the Prevention of Anal Cancer Using Screen and Treat for High-grade Intraepithelial Lesions (IMPACT)
Brief Title: Implementation of Anal Cancer Screening and Treatment in Nigeria
Acronym: IMPACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rebecca Nowak, Assistant Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: HP-00101383; U01CA275053 (NIH)
Record Dates: First submitted 2023-03-14; First posted 2023-04-18 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Education, Medical

STUDY DESIGN:
Intervention Model Description: The way a physician is trained on the detection of HSIL screening and treatment to prevent anal cancer will be modified so that the cancer prevention strategy is readily adopted for a low-to middle-income setting. An implementation science committee will guide the development of the modified training over 3 iterations every 4 months for up to a year. To test if the modified training improves implementation of anal cancer screening and treatment, the physician will first conduct screening after standard training for 12 months. Then the physician will conduct screening after the modified training for 12 months. Depending on the time of when the participants visit the clinic will determine which arm they are enrolled. There is no randomization and the arms are sequential.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Training on screening and treatment of HSIL (e-STH) (Experimental): Tailored training developed to overcome key barriers and promote facilitators unique to implementing HSIL screening and treatment. The development will be driven by the implementation science committee over 3 iterations every 4 months for up to a year to refine the adoption of strategies with the greatest breadth to facilitate implementation.
  Interventions: Behavioral: Enhanced Training on screening and treatment of HSIL (e-STH)
- Standard Screening and treatment of HSIL (No Intervention): The standard screening and treatment of HSIL outlined by the International Anal Neoplasia Society

INTERVENTIONS:
Behavioral: Enhanced Training on screening and treatment of HSIL (e-STH) — Tailored training developed to overcome key barriers and promote facilitators unique to implementing HSIL screening and treatment. The development will be driven by the implementation science committee over 3 iterations every 4 months for up to a year to refine the adoption of strategies with the greatest breadth to facilitate implementation.
  Arms: Enhanced Training on screening and treatment of HSIL (e-STH)

SUMMARY:
The study is a feasibility pilot trial testing 2 types of training protocols on a single physician. The first training protocol is the current standard and was developed in high-income settings. The second training protocol will be developed so tailored to the Nigerian setting. Investigators will test if the physician performs differently in their ability to conduct anal cancer screening and treatment between the 2 training protocols.

DETAILED DESCRIPTION:
In Aim 1, anal cancer screening and treatment based on standard training protocols of how to screen and treat high-grade intraepithelial lesions (HSILs) to prevent anal cancer as developed in high-income settings will be conducted. Investigators will identify barriers and facilitators with learning the procedure with standard training using the Consolidated Framework for Implementation Research (CFIR). In Aim 2, Investigators will identify strategies to modify the standard training to improve learning on a complicated procedure using the Expert Recommendations for Implementing Change (ERIC) framework. An implementation science committee will co-design and develop an enhanced training on Screening and Treatment of HSIL (e-STH) by matching the barriers identified with CFIR with strategies in ERIC. Investigators will then take an iterative improvement approach to test and refine the implementation of the enhanced training intervention to ensure that HSIL screening and treatment is readily adopted and maintained as part of HIV care. In Aim 3 (CLINICAL TRIAL AIM), Investigators will conduct a Hybrid Type 2 trial using an interrupted time series design to monitor and evaluate outcomes along the implementation continuum. The trial will be conducted at a single clinic to minimize variability. The participant (Physician) will have a pre-period of HSIL screening and treatment for 12 months after standard training. Next, investigators will roll out e-STH for 6 months. Then there will be a post-period of screening for 12 months to evaluate the impact of e-STH. Lastly, there will be 6 months of screening and treatment with minimal involvement of the investigative team to evaluate sustainability.

The study will compare e-STH to standard training in proportion of HSIL detected and treated with secondary outcomes evaluating reach, efficacy, implementation, and sustainability.

ELIGIBILITY:
Inclusion Criteria:

1. Possess a medical degree in medical sciences (MBBS or equivalent)
2. At least 2-5 years of experience working with clinical HIV/AIDS community
3. Must be registered with the medical and dental council of Nigeria
4. Possess a current medical practicing license
5. Willing to work with the Sexual Gender Minority Community

Exclusion Criteria:

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in HSIL detection | 12 months and 30 months
  Evaluate change in HSIL detected between the pre and post period (standard vs e-STH)
Change in HSIL treatment | 12 months and 30 months
  Evaluate change in HSIL treated between the pre and post period (standard vs e-STH)

SECONDARY OUTCOMES:
Change in Reach of intended population | 12 months and 30 months
  Change in number screened per number eligible between the pre and post period
Change in Efficacy of conducting HSIL screening and treatment | 12 months and 30 months
  Compare number needed to screen to reach a plateau in the detection of HSIL between the pre and post period
Change in Implementation of HSIL screening and treatment | 12 months and 30 months
  Compare number of biopsies taken per screening between the pre and post period
Change in Maintenance of HSIL screening and treatment | 18 months and 36 months
  Compare number who return for a 12-month screening between the pre and post period

CONTACTS AND LOCATIONS:
Locations (1):
- International Center for Advocacy on Right to Health (ICARH), Abuja, Nigeria